CLINICAL TRIAL: NCT01777711
Title: Exploring Beliefs and Behaviors About Weight Loss in Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Pro00040490
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
Keywords: mental contrasting; weight loss; obese couples; obesity; overweight; planning; health; diet; exercise; physical activity; goal; goal-setting
MeSH Terms: conditions — Obesity; Weight Loss; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Couple condition (Active Comparator): Couples randomized to the couple condition will undergo the experimental manipulations and both partners will complete all study measures. Both members of the couple will be given body mass index (BMI) based on measurements taken during the intervention. Both will complete three surveys on paper and do some prompted planning and goal-setting together regarding weight loss through healthier eating and physical activity.
  Interventions: Behavioral: Mental Contrasting- Couple
- Individual Condition (Active Comparator): Couples randomized to the individual condition will be stratified on gender and one partner, chosen at random, will undergo the experimental manipulations and complete all study surveys while the other will not (heretofore called the active partner vs. the passive partner). The active partner will receive BMI feedback based on measurements taken during the intervention appointment, complete three surveys, and verbally state some goals and plans for weight loss to the passive partner. The passive partner will not complete any study materials or participate in the intervention during the session.
  Interventions: Behavioral: Mental Contrasting- Individual

INTERVENTIONS:
Behavioral: Mental Contrasting- Individual — Investigators will implement the manipulation of mental contrasting/implementation intentions, focusing on the individual. This will entail 3 steps that involve: 1) contrasting of positive future outcomes associated with present conditions that hinder achievement of positive future outcomes (i.e., barriers); 2) strategies to overcome barriers and hence facilitate weight loss; and 3) construction of implementation intentions.
  Arms: Individual Condition
Behavioral: Mental Contrasting- Couple — Investigators will implement the manipulation of mental contrasting/implementation intentions, focusing on the couple. This will entail 3 steps that involve: 1) contrasting of positive future outcomes associated with present conditions that hinder achievement of positive future outcomes (i.e., barriers); 2) strategies to overcome barriers and hence facilitate weight loss; and 3) construction of implementation intentions.
  Arms: Couple condition

SUMMARY:
This study explores among couples in which both members are obese how the use of mental contrasting along with implementation intentions influence intentions and behavior related to weight loss (eating healthy and exercise), actual weight loss, as well as potential reasons (i.e., mediators) why these changes may occur (e.g., social support, changes in beliefs about weight loss, confidence in being able to eat healthy and diet).

DETAILED DESCRIPTION:
This study explores among couples in which both members are obese how the use of mental contrasting along with implementation intentions influence intentions and behaviors related to weight loss (eating healthy and exercise), actual weight loss, as well as potential reasons (i.e., mediators) why these changes may occur (e.g., social support, changes in beliefs about weight loss, confidence in being able to eat healthy and diet). In mental contrasting procedures, people first imagine a desired future (e.g., eating healthy) and then reflect on the current negative reality (e.g., I snack too much). This process makes people aware of changes needed in the present to obtain future positive outcomes, and thus aids in increasing goal commitment and goal pursuit. In implementation intention procedures, individuals form "if-then" statements about how they will enact their goals in their everyday lives. Implementation intentions are highly effective at helping individuals achieve health behavior change. Recent studies suggest that the combined use of mental contrasting and implementation intentions produce more behavior change than either technique alone (e.g., diet) In this study, investigators test whether these procedures vary in their effectiveness when couple members are instructed to focus on themselves versus the relationship, the latter intended to instill a communal coping mindset (i.e., that losing weight is an issue that needs to be addressed as a couple enacted through mutually cooperative behaviors).

ELIGIBILITY:
Inclusion Criteria:

* Married couples or couples living as married
* living in the same household for at least six months
* both members of couple are obese (BMI > 30).
* must be 18 years or older
* can read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
weight loss | one month
  Measure weight loss between baseline and one month visits

SECONDARY OUTCOMES:
dietary changes | one month
  Look at dietary changes in self-report questionnaire.
number of minutes of physical activity | one month
  Measure minutes of physical activity through self-report questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States